CLINICAL TRIAL: NCT02681354
Title: What is the Influence of Dualtask-training With the BioRescue (Analyses and Rehabilitation of Mobility) on Static Balance, Dynamic Balance During Gait and Cognitive-motor Dual Tasks During Gait: A Randomized Controlled Trial
Brief Title: Dual Task Training in Elderly Using the BioRescue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Peter Feys, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2015-PFE-JSP-01
Record Dates: First submitted 2015-07-06; First posted 2016-02-12 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Mild Cognitive Impairment
Keywords: elderly
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A additional BioRescue training (Experimental): Using a playful rehabilitation, BioRescue
  Interventions: Other: Biorescue training
- Regular training (No Intervention)

INTERVENTIONS:
Other: Biorescue training
  Arms: A additional BioRescue training

SUMMARY:
Mild cognitive impairment (MCI) is accompanied by gait and balance problems while dual tasking. During a 6 to 8 weeks training with the BioRescue (virtual reality), institutionalized elderly people with MCI will relearn dual tasks in combination with balance. Afterwards, the transferring effect on gait in general, balance and cognition will be examined.

ELIGIBILITY:
Inclusion Criteria:

* minimum age: 65
* Participants with increased fall-risk (i.e. Timed Up-and-Go Test (TUG) > 20 sec)
* Participants with Mild Cognitive Impairment (MCI) measured by the Montreal Cognitive Assessment (MoCa < 25). MCI: A state of altered cognition, characterized by a decline in one or more cognitive domains, typically including memory while the independence for daily activities remains intact.
* Participants have a positive result on the 'Stops Walking While Talking' test

Exclusion Criteria:

* Diagnosis of Dementia, based on a specialized diagnostic bilan of a doctor-specialist.
* In rehabilitation for a recent injury or recent prothesis of the upper or lower extremities.
* Serious limitations of the lower and or upper limb.
* Not able to walk more than 10 meters independently (walking-aid allowed).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Static balance | day 1
  measured using the BioRescue
Static balance | week 8
  measured using the BioRescue
Dynamic Balance | day 1
  instrumented timed Up-and-Go test
Dynamic Balance | week 8
  instrumented timed Up-and-Go test
instrumented timed Up-and-Go test while dual-tasking | day 1
  instrumented timed Up-and-Go test while dual-tasking
instrumented timed Up-and-Go test while dual-tasking | week 8
  instrumented timed Up-and-Go test while dual-tasking
"stops walking while talking" test | day 1
  "stops walking while talking" test
"stops walking while talking" test | week 8
  "stops walking while talking" test

SECONDARY OUTCOMES:
fall incidence | up to 8 weeks
  The incidence of falls for each participant will be registered in the institution
cognitive function | day 1
  measured by the MOCA (Montreal Cognitive Assesment)
cognitive function | week 8
  measured by the MOCA (Montreal Cognitive Assesment)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University
Locations (2):
- Belgium (2):
  - Hasselt University, Diepenbeek
  - Woon- en zorgcentrum Sint Elisabeth, Hasselt